CLINICAL TRIAL: NCT05917626
Title: Effectiveness and Implementation of a Digital Intervention for Pediatric Chronic Pain Co-designed With Patients
Acronym: Digital SPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Principal Investigator, Rocio de la Vega de Carranza, PhD, "Ramón y Cajal" Researcher; Principal Investigator, University of Malaga
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: PID2021-122885OA-I00
Record Dates: First submitted 2023-05-08; First posted 2023-06-26 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Adolescents; Digital Health; Psychological Intervention; Co-development; Implementation
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: This study will employ a stepped wedge cluster randomized design in which hospitals are randomized sequentially to initiate the intervention. Prior to initiating patient recruitment, each of the 6 hospitals will be randomized to one of two waves in the stepped wedge design. During the non-exposure periods, patients will receive usual care from the hospital.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: * Clinicians referring participants will be unaware of the study phase
  * Outcomes will be assessed with an online survey
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital SPA (Experimental): A psychological intervention for chronic pain in adolescents administered using an app co-created with patients.
  Interventions: Behavioral: Digital SPA
- Usual Care (No Intervention): Participants assigned to this arm will receive usual care from their hospital.

INTERVENTIONS:
Behavioral: Digital SPA — A psychological digital intervention for chronic pain in adolescents, based on evidence-based Acceptance and Commitment Therapy techniques. The intervention will be co-created with patients in a previous phase of the study, so the exact number or format of sessions and content has not been determined yet.
  Arms: Digital SPA

SUMMARY:
Children and adolescents with chronic pain often lack a proper diagnosis and treatment. Research has shown that, if left untreated, it usually doesn't resolve and continues through adulthood.

The goal of this multi-phase study is to co-develop (with patients), test, and implement a smartphone app called "Digital Solution for Pain in Adolescents" (Digital SPA) which can provide pain management resources to children with chronic pain and their parents, preventing future disability.

Participants will: participate in individual and group interviews, respond to questionnaires online and try a smartphone app.

DETAILED DESCRIPTION:
Phase 1) Focus groups with patients, parents and clinicians (n = 5-6 each) will inform about unmet pain care needs, and provide a starting point for co-designing the intervention.

Phase 2) Content creation and usability testing will be based on the results of Phase 1 and the theory-driven development will follow the latest available evidence and the World Health Organization guidelines on the management of chronic pain in children. The intervention will use validated psychological techniques (particularly Cognitive Behavioral Therapy and Acceptance and Commitment Therapy) focused on improving functioning by teaching pain coping skills, such as: relaxation, goal setting, sleep management, behavioral activation, self-management of negative thoughts and emotions, and communication skills.

Phase 3) Effectiveness and Implementation study. Participants (n = 195) will be adolescents 12-17 years old with chronic pain admitted into any of 6 large hospitals in Spain and one of their parents.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents age 12-17 years
* Has had non-oncologic chronic pain for at least 3 months (e.g., abdominal pain, headache or musculoskeletal pain)
* Has Internet access
* One parent is willing to participate (and both give consent for their child to participate)

Exclusion Criteria:

* Diagnosis of a comorbid serious health condition (e.g., cancer)
* Parent or child does not speak or read Spanish
* Active psychosis or suicidal ideation

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 195 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Interference | Pre-treatment (T1), Mid-treatment (T2; 4 weeks after T1), Post-treatment (T3; 8 weeks after T1) and 3-months follow-up (T4; 3 months after T3).
  Spanish version of the Brief Pain Inventory (BPI) short version. Pain intensity scale scores range from from 0 to 10 , with higher scores indicating greater interference. Interference scores range from 0 to 10, with higher scores indicating greater interference.
Global impression of change after treatment | Post-treatment (T3; 8 weeks after T1) and 3-months follow-up (T4; 3 months after T3).
  11-point scale (0 to 10) with higher scores indicating greater impression of change.
Change in the number of visits to the Emergency Room (ER) due to pain | Pre-treatment (T1), Mid-treatment (T2; 4 weeks after T1), Post-treatment (T3; 8 weeks after T1) and 3-months follow-up (T4; 3 months after T3).
  The number of visits to the ER due to pain during the follow-up period (T3 to T4; 3 months) will be compared with the three months before starting treatment (T1).

SECONDARY OUTCOMES:
Change in pain readiness to change | Pre-treatment (T1), Mid-treatment (T2; 4 weeks after T1), Post-treatment (T3; 8 weeks after T1) and 3-months follow-up (T4; 3 months after T3).
  Readiness to adopt a self-management approach to pain. The Spanish version of the Pain Stages of Change Questionnaire for Adolescents (PSoCQ-A). The Questionnaire has three scales: Pre-contemplation, Contemplation, and Action/Maintenance. Each scale is scored in a 1 to 5 Likert scale, with higher scores indicating a higher level of attitudes in that stage of change. The scale with the highest score indicates which stage the respondent is at.
Change in the dose of pain medication taken | Pre-treatment (T1), Mid-treatment (T2; 4 weeks after T1), Post-treatment (T3; 8 weeks after T1) and 3-months follow-up (T4; 3 months after T3).
  The dose (eg. 25 mg per day) of pain medication taken will be recorded.
Change in the type of pain medication taken | Pre-treatment (T1), Mid-treatment (T2; 4 weeks after T1), Post-treatment (T3; 8 weeks after T1) and 3-months follow-up (T4; 3 months after T3).
  The type (e.g. Non-steroid Anti-inflammatory Drugs, opioids) of pain medication taken will be recorded.
Change in Emotional Distress | Pre-treatment (T1), Mid-treatment (T2; 4 weeks after T1), Post-treatment (T3; 8 weeks after T1) and 3-months follow-up (T4; 3 months after T3).
  The Spanish version of the Social Emotional Distress Scale-Secondary (SEDS-S) will be administered to assess general emotional distress (internalizing symptoms such as anxiety and depression) over the past month. The SEDS-S is a 10-item self-report questionnaire; items are rated from 1 ("Not at all true") to 4 ("Very true / Absolutely true"), with higher total scores indicating greater emotional distress.
Change in Functional Disability | Pre-treatment (T1), Mid-treatment (T2; 4 weeks after T1), Post-treatment (T3; 8 weeks after T1) and 3-months follow-up (T4; 3 months after T3).
  Spanish version of CALI-9. Disability in functioning due to pain (activity limitations) is measured through 9 items to evaluate pain-related activity limitations in youth with chronic pain. Scores range from 1 = not very difficult; to 5 = extremely difficult. Higher scores indicating greater interference with children's activities.
Change in Sleep | Pre-treatment (T1), Mid-treatment (T2; 4 weeks after T1), Post-treatment (T3; 8 weeks after T1) and 3-months follow-up (T4; 3 months after T3).
  Sleep quality will be assessed with the Spanish version of the Pittsburgh Sleep Quality Index, validated for adolescents (PSQI). Scores on 7 components range from 0 to 3, and are the summed (global score range 0 to 21, with higher scores indicating worse sleep quality).
  Insomnia will be assessed with the Spanish version of the Adolescent Insomnia Questionnaire (AIQ). Total scores range from 0 to 52 with higher scores indicating more insomnia symptoms.
Change in Pain Self-efficacy | Post-treatment (T3; 8 weeks after T1) and 3-months follow-up (T4; 3 months after T3).
  Pain self-efficacy will be assessed using the Pain Self-Efficacy Questionnaire (PSEQ). The PSEQ is a 10-item self-report measure that evaluates the extent to which individuals feel capable of functioning despite their pain. Items are rated on a 7-point scale from 0 ("not at all confident") to 6 ("completely confident"). Total scores range from 0 to 60, with higher scores indicating greater pain-related self-efficacy.
Psychological Flexibility and Inflexibility Processes | Pre-treatment (T1), Mid-treatment (T2; 4 weeks after T1), Post-treatment (T3; 8 weeks after T1) and 3-months follow-up (T4; 3 months after T3).
  Psychological flexibility and inflexibility will be assessed using the Multidimensional Psychological Flexibility Inventory (MPFI). The MPFI includes subscales capturing both flexibility and inflexibility across six ACT processes. Items are rated on a 1 ("never true") to 6 ("always true") scale. Subscale scores are computed by summing item responses, with higher scores indicating greater levels of the corresponding process (higher flexibility or higher inflexibility). A global index of psychological flexibility will also be measured using the PsyFlex questionnaire. The PsyFlex consists of 6 items rated on a 1 ("very untrue of me") to 5 ("very true of me") scale. Total scores range from 6 to 30, with higher scores indicating greater psychological flexibility.
Satisfaction with treatment | Post-treatment (T3; 8 weeks after T1).
  Usability and satisfaction with the intervention will be assessed using the mHealth App Usability Questionnaire (MAUQ). The MAUQ includes 18 items rated on a 1 ("strongly disagree") to 7 ("strongly agree") scale. Subscales assess ease of use, interface and satisfaction, and usefulness. Higher scores indicate greater usability and satisfaction with the digital intervention.
Adherence to treatment | From the moment the treatment app is downloaded (T1), to the completion of the treatment period (T3). Up to 10 weeks.
  One measure of implementation will be adherence to the online intervention assessed collecting back-end data such as: number of log-ins or number of treatment sections completed.

OTHER OUTCOMES:
Adverse Events (side effects) | Mid-treatment (T2; 4 weeks after T1), Post-treatment (T3; 8 weeks after T1) and 3-months follow-up (T4; 3 months after T3).
  Adverse Events are not expected given the content of the treatment and its non-invasive nature, however, they will be assessed, recorded and controlled for in the analyses

CONTACTS AND LOCATIONS:
Overall Officials: Rocio de la Vega, PhD, Principal Investigator — University of Malaga
Locations (6):
- Spain (6):
  - Hospital Materno Infantil Torrecardenas, Almería, Almería
  - Hospital Sant Joan de Déu, Barcelona, Barcelona
  - Hospital Materno Infantil Virgen de las Nieves, Granada, Granada
  - Hospital infantil del Hospital Universitario La Paz, Madrid, Madrid
  - Hospital General Universitario Santa Lucía, Cartagena, Murcia
  - Hospital Materno Infantil del Hospital Regional Universitario, Málaga, Málaga

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de la Vega R, Serrano-Ibanez ER, Ruiz-Parraga GT, Palermo TM, Wicksell R, Fernandez-Jimenez E, Oliva S, Roldan S, Monfort L, Pelaez MJ, Leyva Carmona M, Ramirez-Maestre C, Lopez-Martinez AE, Miro J, Esteve R. Protocol for a multi-phase, multi-center, real-world, hybrid effectiveness-implementation study of a digital intervention for pediatric chronic pain co-designed with patients (Digital SPA). Digit Health. 2023 Dec 19;9:20552076231219490. doi: 10.1177/20552076231219490. eCollection 2023 Jan-Dec. PMID 38130799
- See also: Project website — https://psicologiadeldolor.es/en/proyectos/en-curso/